CLINICAL TRIAL: NCT01915290
Title: Self Reported Physical Activity vs Objectively Measured Physical Activity and Its Correlation to Maximal Oxygen Uptake in an Elderly Population: an Observational Study
Brief Title: Physical Activity and Its Correlation to Maximal Oxygen Uptake in an Elderly Population
Acronym: Gen100sub2
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: Gen100sub2
Record Dates: First submitted 2013-07-22; First posted 2013-08-02 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Aging
Keywords: physical activity; maximal oxygen uptake
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1600 elderly participants: Norwegian elderly population

SUMMARY:
This is a substudy of the Generation-100 study (NCT01666340). Self reported physical activity versus objectively measured physical activity and its correlation to maximal oxygen uptake in an elderly Norwegian population (observational study).

DETAILED DESCRIPTION:
Data is collected using activity monitors. This data then compared to self reported physical activity obtained through questionnaires. Questionnaires are based on recall. Overall physical activity will then be correlated to maximal oxygen uptake to see whether people with high activity also have high maximal oxygen uptake.

ELIGIBILITY:
Inclusion Criteria:

* ability to walk at least 1km,
* born in 1938,1939,1940,1941 or 1942
* Sufficiently good health to be able to take part in the study, as determined by the researchers

Exclusion Criteria:

* Illness or disability that precludes exercise or hinders completion of the study
* Uncontrolled hypertension
* Symptomatic valve disease, hyper tropic cardio-myopathy or unstable angina
* Active cancer
* Test results indicating that study participation is unsafe
* Inclusion in other studies conflicting with participation in this one

Ages: 70 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Norwegian elderly population 70-77 years of age
Sampling Method: Non-Probability Sample
Enrollment: 1237 (Actual)
Dates: Start 2012-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Correlation between maximal oxygen uptake and activity level | baseline
  maximal oxygen uptake measured using Metamax on a Treadmill. Activity level assessed using triaxial activity monitors.

SECONDARY OUTCOMES:
Difference between self reported recall physical activity and activity monitor measured physical activity | Baseline
  self reported Physical Activity is assessed by having participants fill out a questionnaire (developed by HUNT) outlining their Physical Activity (through recall).
  Physical activity is objectively measured using triaxial accelerometers.

OTHER OUTCOMES:
total daily energy expenditure | Baseline
  Measured through triaxial accelerometer.
activity energy expenditure | baseline
  Measured using triaxial accelerometer
sedentary time | baseline
  Measured using triaxial accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Dorthe Stensvold, PhD, Principal Investigator — Norwegian University of Science and Technology; Ulrik Wisløff, PhD, Study Chair — Norwegian University of Science and Technology